CLINICAL TRIAL: NCT04917419
Title: Prise en Charge infirmière Des Anomalies du Sommeil et du Rythme Circadien Par luminothérapie et/ou un Programme Court de psychoéducation Chez Des Patients Souffrant de Troubles Bipolaires
Brief Title: Nursing Care of Bipolar Patients With Sleeping Disorders Using Luminotherapy and /or Psychoeducation Program (BIPLUMINO)
Acronym: BIPLUMINO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A02526-33
Record Dates: First submitted 2021-02-26; First posted 2021-06-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luminotherapy and Psychoeducation Program (Experimental)
  Interventions: Other: Luminotherapy and /or Psychoeducation Program
- Psychoeducation Program (Active Comparator)
  Interventions: Other: Luminotherapy and /or Psychoeducation Program

INTERVENTIONS:
Other: Luminotherapy and /or Psychoeducation Program — TO complete

SUMMARY:
Bipolar disorder affects more than 1% of the population. This pathology is considered as one of the most serious psychiatric disorder because of it is high suicide rates. It impacts patients life quality on many aspects, and specially their sleeping and circadian Rhythms. This can lead to more severe symptoms up to for thymic relapses. It was shown that Luminotherapy and Psychoeducation Program have a positive impact on these type of symptoms.

ELIGIBILITY:
Main inclusion Criteria:

* Bipolar disorder (type 1 and 2 according to DSM V)
* Mood Disorder Questionnaire MDQ ˂ 7
* Sleeping and Circadian Rhythms Disorders
* Under treatment

Main exclusion Criteria:

* No addiction except for tobacco
* Narcolepsy
* Sleep Apnea
* Psychiatric comorbidities
* Suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of days in-hospital | Day 0 to Day 365
  Number of days patients spent in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No